CLINICAL TRIAL: NCT05352945
Title: Effectiveness of HYPNOsis Masks in the Management of Pain and Anxiety During Botulinum TOXin Injections in the Treatment of Idiopathic Overactive Bladder: a Multicenter Randomized Parallel Group Study.
Brief Title: Effectiveness of HYPNOsis Masks During Botulinum TOXin Injections in Idiopathic Overactive Bladder(HypnoTox)
Acronym: HypnoTox
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insuffisant patient recruyting
Sponsor: Centre Hospitalier de Roubaix (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-004
Record Dates: First submitted 2022-04-25; First posted 2022-04-29 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Idiopathic Overactive Bladder
Keywords: hypnosis mask; idiopathic overactive bladder; pain; anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Patients newly eligible for treatment of idiopathic overactive bladder with botulinum toxin injection will be randomised into two groups before injection:
  * Group 1: conventional anaesthesia
  * Group 2: conventional anaesthesia and use of self-hypnosis mask
Masking Description: Blinding is not possible with the self-hypnosis mask as it emits sounds and lights for its effect.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control arm (No Intervention): conventional anaesthesia
  The botulinum toxin injection procedure will be carried out in the standard way, according to the recommendations applicable in France, and after local anaesthesia.
- interventional arm (Experimental): conventional anaethesia and use of the self-hypnosis mask
  The mask and the helmet are positioned and activated 10 minutes before the procedure, with the "travel to india" programme chosen because it was developed for pain management and its duration is compatible with the procedure (25 minutes).
  Interventions: Device: HyPNOS self-hypnosis mask from DREAMINZZ

INTERVENTIONS:
Device: HyPNOS self-hypnosis mask from DREAMINZZ — The use of the HyPNOS self-hypnosis mask from DREAMINZZ allows patients to immerse themselves in a state of self-hypnosis.
  A Hypnos session is a narrative accompanied by spatialized sounds (3D) and ambiance for an immersive experience.
  We aim to evaluate the use of the HyPNOS mask in the management of pain and anxiety in botulinum toxin injections
  Arms: interventional arm

SUMMARY:
Monocenter, prospective, randomized, parallel group study (1:1) evaluating the efficacy of self-hypnosis performed by mask on pain and anxiety in patients receiving botulinum toxin injections in the treatment of idiopathic overactive bladder refractory to conventional pharmacological treatment.

Patients will be randomized into two groups before injection:

* Group 1: conventional anesthesia
* Group 2: conventional anesthesia and use of the self-hypnosis mask

At the end of the procedure, the patient will express the pain felt thanks to the VAS (Visual Analog Scale) and will answer a questionnaire of anxiety (STATE-TRAIT Anxiety Inventory).

DETAILED DESCRIPTION:
Day 0: 1st consultation for overactive bladder refractory to drug treatment: verification of inclusion and non-inclusion criteria. Proposal of the study to the patient and handing over of the information note relating to the study.

D15: Collection of consent and randomisation - execution of the procedure

Botulinum toxin injection procedure

Control arm: conventional anaesthesia The botulinum toxin injection procedure will be carried out in a standard manner, according to French guidances, and after local anaesthesia as specified below.

For the procedure, the patient will be hospitalised in a urological day hospital. She must have a sterile cytobacteriological exam of urine 10 days before the procedure or be on antibiotics, and must not have any coagulation problems.

A local anaesthetic is given 30 minutes before the procedure according national guidances.

Experimental arm: conventional anaesthesia and use of the self-hypnosis mask

Same procedure as described for the control arm with the addition of the self-hypnosis mask during the procedure:

The mask and the headphones are positioned and activated 10 minutes before the procedure, with the program "travel to India" chosen because it was developed for pain management and of a duration compatible with the procedure (25 minutes).

A short presentation acting as a pre-hypnotic speech can introduce the use of the mask on a patient in order to orientate the effects in the desired goal (analgesia, relaxation, etc.).

After connecting the mask to the mobile application, the caregiver will set the appropriate program for the treatment, place the mask over the patient's closed eyes, place the headphones over the patient's ears as well and start the session in question.

Following the procedure, monitoring in the day hospital and evaluation at 30 minutes of the procedure by a trained nurse, of the pain felt during the insertion of the cystoscope and during the injections by VAS.

Completion of the STATE-TRAIT Anxiety Inventory test.

D45: Regular monitoring consultation with evaluation of treatment effectiveness. Collection of data concerning complications (haematuria, urine retention and urinary tract infection). Discharge from the study.

ELIGIBILITY:
Inclusion Criteria:

* Woman with non-neurological overactive bladder, confirmed by urodynamic assessment and cystoscopy, having resisted a well-conducted pharmacological treatment (trials of various anticholinergics).
* Age over 18 years
* Having understood the study and agreed to participate (signing of informed consent)
* Beneficiary of a health insurance plan

Exclusion Criteria:

* Neurological patient: tetraplegic, paraplegic, multiple sclerosis for a reliable pain assessment
* Patients who have already been injected with botulinum toxin in the treatment of this pathology.
* Psychiatric pathology at risk of decompensation with self-hypnosis
* Patients who are difficult to assess because of a psychological disorder that does not allow them to answer questionnaires and pain assessment scales
* Patients under court protection, guardianship or curatorship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-11-25 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
Pain felt at the time of the injections | During the botulinum toxin injections
  Measured by a Visual Analogue Scale (VAS) rated from 0 to 100 millimetres

SECONDARY OUTCOMES:
Anxiety | During the botulinum toxin injections
  Measured by the STAI Forme Y-A which assesses the state of anxiety at a given time
Pain felt on insertion of the cystoscope | During insertion of the cystoscope
  Measured by a Visual Analogue Scale (VAS) rated from 0 to 100 millimetres
Occurrence of complications | During the 7 days post-procedure
  Hematuria, Acute Urine Retention and Urinary Tract Infection
Success of the 50IU procedure | At 1 month post-procedure
  Assessed by the doctor

CONTACTS AND LOCATIONS:
Overall Officials: François Pecoux, Doctor, Principal Investigator — CH ROUBAIX
Locations (1):
- CH de Roubaix, Roubaix, France

IPD SHARING:
Plan to Share IPD: No
The database created will remain the property of the Hospital Center of Roubaix. The Hospital Center of Roubaix will carry out the main publication of the research.
  Once this has been done, the investigating centres that participated in the research can request access to the database for the purpose of secondary publications.
  If the request is successful, the database will be transmitted securely and completely anonymously to the applicant.

REFERENCES:
- [Background] Zhang ZS, Wang XL, Xu CL, Zhang C, Cao Z, Xu WD, Wei RC, Sun YH. Music reduces panic: an initial study of listening to preferred music improves male patient discomfort and anxiety during flexible cystoscopy. J Endourol. 2014 Jun;28(6):739-44. doi: 10.1089/end.2013.0705. Epub 2014 Mar 31. PMID 24548148
- [Result] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Int Urogynecol J. 2010 Jan;21(1):5-26. doi: 10.1007/s00192-009-0976-9. Epub 2009 Nov 25. PMID 19937315
- [Result] Game X, Karsenty G, Ruffion A, Amarenco G, Ballanger P, Chartier-Kastler E, Cosson M, Costa P, Fatton B, Deffieux X, Haab F, Hermieu JF, Le Normand L, Saussine C, Denys P. [Idiopathic overactive bladder and BOTOX((R)): Literature review]. Prog Urol. 2015 Jun;25(8):461-73. doi: 10.1016/j.purol.2015.01.006. Epub 2015 Feb 3. French. PMID 25662706
- [Result] Milsom I, Abrams P, Cardozo L, Roberts RG, Thuroff J, Wein AJ. How widespread are the symptoms of an overactive bladder and how are they managed? A population-based prevalence study. BJU Int. 2001 Jun;87(9):760-6. doi: 10.1046/j.1464-410x.2001.02228.x. PMID 11412210
- [Result] Coyne KS, Sexton CC, Kopp ZS, Ebel-Bitoun C, Milsom I, Chapple C. The impact of overactive bladder on mental health, work productivity and health-related quality of life in the UK and Sweden: results from EpiLUTS. BJU Int. 2011 Nov;108(9):1459-71. doi: 10.1111/j.1464-410X.2010.10013.x. Epub 2011 Mar 3. PMID 21371240
- [Result] Denys P, Le Normand L, Ghout I, Costa P, Chartier-Kastler E, Grise P, Hermieu JF, Amarenco G, Karsenty G, Saussine C, Barbot F; VESITOX study group in France. Efficacy and safety of low doses of onabotulinumtoxinA for the treatment of refractory idiopathic overactive bladder: a multicentre, double-blind, randomised, placebo-controlled dose-ranging study. Eur Urol. 2012 Mar;61(3):520-9. doi: 10.1016/j.eururo.2011.10.028. Epub 2011 Oct 25. PMID 22036776
- [Result] Schurch B, Schmid DM, Stohrer M. Treatment of neurogenic incontinence with botulinum toxin A. N Engl J Med. 2000 Mar 2;342(9):665. doi: 10.1056/NEJM200003023420918. No abstract available. PMID 10702067
- [Result] Karsenty G, Baverstock R, Carlson K, Diaz DC, Cruz F, Dmochowski R, Fulford S, Giannantoni A, Heesakkers J, Kaufmann A, Peyrat L, Thavaseelan J, Dasgupta P. Technical aspects of botulinum toxin type A injection in the bladder to treat urinary incontinence: reviewing the procedure. Int J Clin Pract. 2014 Jun;68(6):731-42. doi: 10.1111/ijcp.12360. Epub 2014 Jan 29. PMID 24472109
- [Result] Hermieu JF, Ballanger P, Amarenco G, Chartier-Kastler E, Cosson M, Costa P, Fatton B, Deffieux X, Denys P, Game X, Haab F, Karsenty G, Le Normand L, Ruffion A, Saussine C. [Guidelines for practical usage of botulinum toxin type A (BoNTA) for refractory idiopathic overactive bladder management]. Prog Urol. 2013 Dec;23(17):1457-63. doi: 10.1016/j.purol.2013.10.006. Epub 2013 Nov 7. French. PMID 24286546
- [Result] Kendrick C, Sliwinski J, Yu Y, Johnson A, Fisher W, Kekecs Z, Elkins G. Hypnosis for Acute Procedural Pain: A Critical Review. Int J Clin Exp Hypn. 2016;64(1):75-115. doi: 10.1080/00207144.2015.1099405. PMID 26599994
- [Result] Noergaard MW, Hakonsen SJ, Bjerrum M, Pedersen PU. The effectiveness of hypnotic analgesia in the management of procedural pain in minimally invasive procedures: A systematic review and meta-analysis. J Clin Nurs. 2019 Dec;28(23-24):4207-4224. doi: 10.1111/jocn.15025. Epub 2019 Sep 3. PMID 31410922
- [Result] Gezginci E, Iyigun E, Kibar Y, Bedir S. Three Distraction Methods for Pain Reduction During Cystoscopy: A Randomized Controlled Trial Evaluating the Effects on Pain, Anxiety, and Satisfaction. J Endourol. 2018 Nov;32(11):1078-1084. doi: 10.1089/end.2018.0491. PMID 30280915